CLINICAL TRIAL: NCT04521257
Title: Development of Urdu Version of Short Form 36 Health Questionnaire; Validation and Reliability Analysis in Healthy Population
Brief Title: Development of Urdu Version of Short Form 36 Health Questionnaire
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/20/2027 Shaheer Haider
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Quality of Life
Keywords: Health Related Quality of Life; Public Health; Health Status Indicators

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Quality of life (QOL) is an overarching term for the quality of the various domains in life. It is a standard level that consists of the expectations of an individual or society for a good life. These expectations are guided by the values, goals and socio-cultural context in which an individual lives. It is a subjective, multidimensional concept that defines a standard level for emotional, physical, material and social well-being. The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and an abbreviated variant of it, the SF-6D, is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. The original SF-36 stemmed from the Medical Outcome Study, MOS, which was conducted by the RAND Corporation. The primary objectives of this research were to translate, validate and generate normative data on the SF-36 health survey for using among Urdu speaking residents of Pakistan.SF-36 health questionnaire is first translated into Urdu and then apply on healthy subjects to check the validity and reliability of this scale . Instrument will be first translated from English to Urdu by two experts. Both these experts were fluent in English and Urdu language. One expert belongs to allied health care profession and other expert will be junior life scientist. The third expert compares the initial to Urdu translation and formulated the first draft of SF-36 Health Questionnaire. Content validity of SF-36 Health Questionnaire was established by committee method. 10 experts from physical therapy field rate the all 36 items of the SF-36 Health Questionnaire on content validity index developed by RAND Corporation. They rate each item of SF-36 Health Questionnaire for its relevance, clarity, simplicity, and ambiguity on four point ordinal likert scale. Data will be analyzed using SPSS v 25. Intra class correlation coefficient, chronbach alpha and factor analysis will be used to analyses the data.

DETAILED DESCRIPTION:
The 36-item Short Form Health Survey is a brief self administered questionnaire that generates scores across eight dimensions of health: physical functioning (PF), role limitations due to physical problems (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), mental health (MH), and one single item scale on health transition. It has proved useful in monitoring population health, estimating the burden of different diseases, monitoring outcomes in clinical practice, and evaluating treatment effects. The improved longevity suggests that health status can no longer be well assessed by population mortality statistics; there is a consensus to view health in terms of people's subjective assessment of wellbeing and ability to perform social roles the centrality of people's point of view in monitoring health related quality of life has led to the proliferation of instruments and a rapid development of theoretical literature. Interest in measuring the aspects of health most closely related to quality of life usually referred to as health-related. Quality of life (HR-QOL) has increased in recent years in Pakistan as in other countries. Advances have been made in methods for describing patients' subjective health status using standardized measures, and several valid and reliable patient- based measures are available either as generic or disease and treatment targeted questionnaires. However, most of these are in English and are intended for use in English-speaking settings.With few but relevant exceptions that were actually translated or developed as part of Multilanguage and multinational projects. Most of such efforts were produced by isolated groups of researchers who seldom published their findings in peer-reviewed journals. Among the so-called generic measures, the MOS 36- Item Short Form Health Survey (SF-36) is known for its comprehensiveness, brevity, and high standards of reliability and validity. It was first translated by independent Italian teams in 1990. With the launch of the International Quality of Life Assessment (IQOLA) project. The reliability and validity of the SF-36 have been well documented by the developers of the instrument. A comparison of a series of generic health status measures indicated that the SF-36 is not only psychometrically sound but is also more responsive to clinical improvement than the other instruments tested. Moreover, health functioning changed in the hypothesized direction with increased age, socioeconomic status and disease status in a population-based longitudinal study of the SF-36, which suggests that the instrument is sensitive to changes in the health of the general population. The SF-36 has been cross- culturally translated and Adapted to many cultures and languages. To the Author's knowledge, there is no version of SF-36 in Urdu. Lack of Urdu version of the SF-36 impedes comparison of interventions performed in Urdu rehabilitation clinics with those performed elsewhere.

ELIGIBILITY:
Inclusion Criteria:

Age between 20 to 60 years both male and female subjects

Exclusion Criteria:

Current health problems such as chronic allergy, back pain, visual impairments, chronic skin problems, chronic lung problems, deafness or hearing problems, functional impairment in leg or arm or other chronic health problems

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy subjects aged between 20 to 60 years both male and female subjects will be included.Current health problems such as chronic allergy, back pain, visual impairments, chronic skin problems, chronic lung problems, deafness or hearing problems, functional impairment in leg or arm or other chronic health problems
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Short Form 36 | 2nd Day
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Riphah Rehabiliation Clinic, Lahore, Punjab Province
  - Riphah International University, Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Background] Kolotkin RL, Andersen JR. A systematic review of reviews: exploring the relationship between obesity, weight loss and health-related quality of life. Clin Obes. 2017 Oct;7(5):273-289. doi: 10.1111/cob.12203. Epub 2017 Jul 10. PMID 28695722
- [Background] Puciato D, Rozpara M, Borysiuk Z. Physical Activity as a Determinant of Quality of Life in Working-Age People in Wroclaw, Poland. Int J Environ Res Public Health. 2018 Mar 29;15(4):623. doi: 10.3390/ijerph15040623. PMID 29596312
- [Background] Hasanvand S, Rassouli M, Mandegari Z, Salmani N, Moghimkhan F. A Critical Review of Instruments Measuring the Quality of Life of Cancer Patients in Iranian Studies and Their Psychometrics Properties. Asian Pac J Cancer Prev. 2019 Feb 26;20(2):333-343. doi: 10.31557/APJCP.2019.20.2.333. PMID 30803191
- [Background] Lu WC, Tzeng NS, Kao YC, Yeh CB, Kuo TB, Chang CC, Chang HA. Correlation between health-related quality of life in the physical domain and heart rate variability in asymptomatic adults. Health Qual Life Outcomes. 2016 Oct 21;14(1):149. doi: 10.1186/s12955-016-0555-y. PMID 27765048